CLINICAL TRIAL: NCT04511819
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Losmapimod in Adult Subjects With COVID-19 (LOSVID STUDY)
Brief Title: Losmapimod Safety and Efficacy in COVID-19
Acronym: LOSVID
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to the rapidly evolving environment for the treatment of Covid-19 and ongoing challenges to identify and enroll qualified patients to participate.
Sponsor: Fulcrum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIS-001-2020
Record Dates: First submitted 2020-08-08; First posted 2020-08-13 (Actual); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
Keywords: COVID-19 pandemic; COVID-19 virus disease; COVID-19 virus infection; SARS-CoV-2 infection; coronavirus disease 2019; 2019 novel coronavirus disease; 2019 novel coronavirus infection
MeSH Terms: conditions — COVID-19 | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Intervention Model Description: This study is a randomized, double-blind, placebo-controlled study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be performed in a double-blind fashion. The investigator, study staff, subjects, Sponsor, and monitor will remain blinded to the treatment until study closure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Losmapimod (Experimental): COVID-19 patients with PCR confirmation will receive Losmapimod 15 mg twice daily given as two 7.5 mg tablets per dose by mouth; for a total of 4 pills or 30 mg daily for 14 days.
  Interventions: Drug: Losmapimod oral tablet
- Placebo (Placebo Comparator): COVID-19 patients with PCR confirmation will receive Placebo twice daily given as two tablets per dose by mouth; for a total of 4 tablets daily for 14 days.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Losmapimod oral tablet — Losmapimod will be administered with food when possible.
  Arms: Losmapimod
Drug: Placebo oral tablet — Placebo will be administered with food when possible.
  Arms: Placebo

SUMMARY:
The therapeutic hypothesis for the use of losmapimod in COVID-19 disease is that increased mortality and severe disease is caused by p38 mitogen-activated protein kinase (MAPK)-mediated exaggerated acute inflammatory response resulting from SARS-CoV-2 infection.

The study Sponsor hypothesizes that the early initiation of p38α/β inhibitor therapy in patients hospitalized with moderate COVID-19 who are at increased risk of a poor prognosis based on older age and elevated systemic inflammation will reduce clinical deterioration including progression to respiratory failure and death.

To address this hypothesis, Fulcrum Therapeutics is conducting a Phase 3, multicenter, randomized, double-blind, placebo-controlled study that will evaluate the safety and efficacy of losmapimod versus placebo in subjects 40 and older who are hospitalized with moderate COVID-19 disease.

DETAILED DESCRIPTION:
The therapeutic hypothesis for the use of losmapimod in COVID-19 disease is that increased disease severity and consequent increased mortality is caused by p38 mitogen-activated protein kinase (MAPK)-mediated exaggerated acute inflammatory response resulting from SARS-CoV-2 infection.

It is anticipated that the early initiation of p38α/β inhibitor therapy in patients with moderate COVID-19 will prevent further clinical deterioration and reduce the need for both increased respiratory support as well as mortality. This is the main hypothesis for this study.

To address this hypothesis, Fulcrum Therapeutics is conducting a Phase 3, multicenter, randomized, double-blind, placebo-controlled study that will evaluate the safety and efficacy of losmapimod versus placebo in subjects with COVID-19 disease.

Losmapimod is currently in Phase 2 clinical trials for the treatment of facioscapulohumeral dystrophy (FSHD) and has previously been administered to more than 3600 adult healthy volunteers and subjects including participants in a large Phase 3 trial which evaluated clinical outcomes and safety after major cardiovascular events.

Patients will participate in this study for approximately 34 days. The total treatment duration will be 14 days. Subjects will be evaluated during a 3 day pre-treatment period (Screening and Baseline Visits) to establish pre-treatment baseline assessments and eligibility. Subjects will then be randomized to treatment with losmapimod or placebo for 14 days and assessed frequently for changes from pre-treatment in various clinical outcome assessments. Patients must have a confirmed diagnosis of COVID-19 by viral PCR prior to randomization and first dosing. Patients will receive 15 mg of losmapimod, or placebo twice daily given as two 7.5 mg tablets per dose by mouth: for a total of 4 pills or 30 mg daily for 14 consecutive days. All study visits during the first week of treatment are anticipated to be conducted in the inpatient setting while later visits are anticipated to be conducted as outpatient.

The primary endpoint of the study is to assess the efficacy of losmapimod tablets compared with placebo for the treatment of COVID-19 when administered concurrently with the local standard of care. Secondary endpoints include evaluating the effect of losmapimod compared with placebo on clinical outcomes, clinical status, effect on survival, safety, and tolerability and to characterize changes in the levels of SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide written informed consent
* Willing and able to comply with all study procedures.
* Confirmed infection with SARS-CoV-2 virus at or before the baseline visit by polymerase chain reaction (PCR) testing
* ≤7 days to the time of randomization from the time of collection of the specimen that tested positive for the SARS-CoV-2 virus
* Hospitalization at the time of the baseline visit
* ≥90% oxygen saturation on room air and/or ≥94% oxygen saturation on oxygen administration at 2 L/min by nasal cannula at the baseline visit
* Radiographic (X-ray or computed tomography scan, per local standard of care) and/or clinical evidence of pulmonary involvement consistent with COVID-19 at screening or baseline, per the judgment of the investigator
* Clinical syndrome consistent with COVID-19 at screening, per the judgment of the investigator (CDC 2020)
* CRP at screening >15 mg/L (i.e., >1.5 mg/dL) on local laboratory testing
* Agrees to practice an approved method of birth control

Exclusion Criteria:

* Inability to take oral medication at screening or baseline visit
* Evidence at screening or baseline of critical COVID-19 disease (e.g., cardiac failure, septic shock) or severe pulmonary involvement)
* Positive pregnancy test at screening for women of childbearing potential
* Lactating female at baseline for women of childbearing potential Note: A female will be considered eligible who is lactating at screening if she agrees to discontinue breastfeeding for the duration of the trial plus 14 days post last dose
* ≥5 × upper limit of normal (ULN) for alanine or aspartate aminotransferases or total bilirubin >1.5 × ULN at screening or known history of Child-Pugh Class C, hepatitis B or C, or HIV infection
* Glomerular filtration rate <30 mL/min/1.73 m2 at screening
* QTcF >450 msec for male or >470 msec for females or evidence of cardiac dysrhythmia at screening
* Significant history or evidence of clinically significant disorder, condition, current illness, illicit drug or other addiction, or disease that, in the opinion of the Investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion
* Has been treated with immunomodulators or immunosuppressants including, but not limited to, interleukin (IL)-6 inhibitors, tumor necrosis factor (TNF) inhibitors, anti-IL-1 agents, and Janus kinase inhibitors, within 5 half-lives or 30 days, whichever is longer, prior to randomization, or plan to receive these agents any time during the study period
* Treatment with hydroxychloroquine/ chloroquine in the past 30 days or plan to receive these agents as part of investigational clinical trials or SOC any time during the study period
* Recent (within 30 days) or current participation in other COVID-19 therapeutic trials or expanded access programs
* Prior or current participation in COVID-19 vaccine trials

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Ziegler, MD, FASA, Study Director — Fulcrum Therapeutics
Locations (16):
- United States (7):
  - University of California Irvine - Irvine Medical Center, Irvine, California
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Memorial Hermann Hospital South West, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - United Medical Memorial Hospital, Houston, Texas
- Brazil (4):
  - Hospital Universitario Cassiano Antonio de Moraes-HUCAM/Hospital das Clinicas, Vitória, Espírito Santo
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Irmandade de Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Santa Catarina
  - Hospital Santa Paula, São Paulo, São Paulo
- Mexico (4):
  - Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco
  - Nuevo Hospital Civil de Guadalajara, Guadalajara, JC
  - JM Research Cuernavaca, Cuernavaca, Morelos
  - Centro para el Desarrollo de la Medicina y de Asistencia Médica Especializada, S.C., Culiacán, Sinaloa
- Hospital Nacional Carlos Alberto Seguín Escobedo - EsSalud Arequipa, Arequipa, AR, Peru

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grimes JM, Grimes KV. p38 MAPK inhibition: A promising therapeutic approach for COVID-19. J Mol Cell Cardiol. 2020 Jul;144:63-65. doi: 10.1016/j.yjmcc.2020.05.007. Epub 2020 May 16. PMID 32422320
- [Background] Jimenez-Guardeno JM, Nieto-Torres JL, DeDiego ML, Regla-Nava JA, Fernandez-Delgado R, Castano-Rodriguez C, Enjuanes L. The PDZ-binding motif of severe acute respiratory syndrome coronavirus envelope protein is a determinant of viral pathogenesis. PLoS Pathog. 2014 Aug 14;10(8):e1004320. doi: 10.1371/journal.ppat.1004320. eCollection 2014 Aug. PMID 25122212
- [Background] Vukmanovic-Stejic M, Chambers ES, Suarez-Farinas M, Sandhu D, Fuentes-Duculan J, Patel N, Agius E, Lacy KE, Turner CT, Larbi A, Birault V, Noursadeghi M, Mabbott NA, Rustin MHA, Krueger JG, Akbar AN. Enhancement of cutaneous immunity during aging by blocking p38 mitogen-activated protein (MAP) kinase-induced inflammation. J Allergy Clin Immunol. 2018 Sep;142(3):844-856. doi: 10.1016/j.jaci.2017.10.032. Epub 2017 Nov 17. PMID 29155150
- [Background] Watz H, Barnacle H, Hartley BF, Chan R. Efficacy and safety of the p38 MAPK inhibitor losmapimod for patients with chronic obstructive pulmonary disease: a randomised, double-blind, placebo-controlled trial. Lancet Respir Med. 2014 Jan;2(1):63-72. doi: 10.1016/S2213-2600(13)70200-5. Epub 2013 Dec 5. PMID 24461903
- [Background] World Health Organization (WHO). WHO R&D blueprint novel coronavirus COVID-19 therapeutic trial synopsis. Draft Feb 18, 2020.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 5 sites in the United States and 3 sites in Brazil.
Pre-assignment Details: This was a Phase 3, multicenter, randomized, double-blind, placebo-controlled study which evaluated the safety and efficacy of losmapimod versus placebo on a background of standard of care in participants with Coronavirus disease-2019 (COVID-19) disease (LOSVID Study)
Groups:
- Placebo: Participants were randomized to receive matching placebo tablets orally (PO) twice per day (BID) with food whenever possible and with 240 milliliters (mL) of room temperature water for 14 days.
- Losmapimod 15 Milligrams (mg): Participants were randomized to receive losmapimod tablets 15 mg (2×7.5 mg tablets/dose) PO BID with food whenever possible and with 240 mL of room temperature water for 14 days.
Period: Overall Study
Arm/Group | Placebo | Losmapimod 15 Milligrams (mg)
Started | 26 | 22
Completed | 20 | 17
Not Completed | 6 | 5
Not completed — Non-compliance with study drug | 5 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Protocol deviation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: included all participants who were randomized and received any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Losmapimod 15 Milligrams (mg) | Total
Number analyzed (Participants) | 26 | 22 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.7 (12.15) | 60.8 (10.00) | 59.1 (11.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 15 | 13 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 16 | 38
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 19 | 12 | 31
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Progressed to Death or Respiratory Failure by Day 28
Description: Respiratory failure was defined as either need for mechanical ventilation (invasive or non-invasive) or high flow oxygen (defined by greater than 15 liters per minute [LPM] flow of oxygen to maintain oxygen saturation between 90% and 95%), sustained for at least 48 hours, at any time during the study. The fitted logistic regression model was used to predict the response rate for every participant in the study who had received the treatment or the control intervention. The efficacy of Losmapimod was assessed by the development of progression to critical disease as evidence of mortality or development of respiratory failure by Day 28. Percentage of participants who progressed to death or respiratory failure by Day 28 has been presented.
Time Frame: Up to Day 28
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Losmapimod 15 Milligrams (mg)
Number analyzed (Participants) | 26 | 22
Percentage of participants | 61.5 | 75.0
Statistical Analysis 1: Comparison: Placebo vs Losmapimod 15 Milligrams (mg); Test type: Other; p = 0.8762, Regression, Logistic; Risk Difference (RD) = -0.087, 95% CI 2-sided [-0.347 to 0.174]

2. Secondary Outcome: Change From Baseline in Clinical Status at Days 7 and 14 Assessed on the 9-point World Health Organization (WHO) Ordinal Scale
Description: Change in clinical status between Baseline and at Days 7 and 14 was modeled using ordinal logistic regression models, adjusting for stratification factors, sex and baseline C-reactive protein (CRP). WHO 9-point ordinal scale included score ranges as: 0:No clinical evidence of the disease, 1: Discharged from the hospital and without any limitation, 2: Discharged from the hospital but with limitation of activities, 3: Hospitalized but not requiring oxygen therapy, 4: Oxygen therapy but not requiring high-flow or non-invasive ventilation, 5: Noninvasive ventilation or high-flow oxygen therapy, 6: Intubation and mechanical ventilation, 7: Ventilation plus additional organ support and 8: Death. Higher scores indicated worse clinical status. Baseline was defined as the last measurement prior to the first dose of study drug. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and at Day 7 and Day 14
Population: Full Analysis Set. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Losmapimod 15 Milligrams (mg)
Number analyzed (Participants) | 25 | 22
Scores on a scale
  Day 7: number analyzed (Participants) | 24 | 18
  Day 7 | -1.6 (1.14) | -1.4 (1.58)
  Day 14 | -2.2 (0.83) | -2.0 (1.31)

3. Secondary Outcome: Total Number of Study Days Free of Oxygen Supplementation
Description: A Poisson regression model or a negative binomial model was used to assess the relationship with treatment, adjusting for stratification factors, sex, baseline CRP and number of days on study (as applicable). Total number of study days free of oxygen supplementation has been presented.
Time Frame: Up to Day 28
Population: Full Analysis Set. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Losmapimod 15 Milligrams (mg)
Number analyzed (Participants) | 26 | 18
Days | 24.0 (3.52) | 20.6 (8.80)

4. Secondary Outcome: Percentage of Participants Reporting All-cause Mortality at Day 28
Description: Percentage of participants who reported death have been presented.
Time Frame: At Day 28
Population: Full Analysis Set. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Losmapimod 15 Milligrams (mg)
Number analyzed (Participants) | 24 | 16
Percentage of participants | 0.0 | 0.0

5. Secondary Outcome: Number of Study Days Alive
Description: A Poisson regression model or a negative binomial model was used to assess the relationship with treatment, adjusting for stratification factors, sex, baseline CRP and number of days on study (as applicable). Number of study days alive has been presented.
Time Frame: Up to Day 28
Population: Full Analysis Set. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Losmapimod 15 Milligrams (mg)
Number analyzed (Participants) | 26 | 18
Days | 27.9 (0.27) | 27.8 (0.51)

6. Secondary Outcome: Number of Participants Reporting Non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment. Number of participants with non-serious AEs and SAEs has been presented.
Time Frame: Up to Day 28
Population: Safety Analysis Set: included all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Losmapimod 15 Milligrams (mg)
Number analyzed (Participants) | 26 | 22
Participants
  Non-serious AEs | 15 | 12
  SAEs | 0 | 4

ADVERSE EVENTS:
Time Frame: Up to Day 28
Description: Safety population which included all participants who received any study drug.
Arm/Group | Placebo | Losmapimod 15 Milligrams (mg)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/26 | 4/22
Other Adverse Events (participants affected / at risk) | 15/26 | 12/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=26) | Losmapimod 15 Milligrams (mg) (N=22)
Atrial fibrillation (Cardiac disorders) | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=26) | Losmapimod 15 Milligrams (mg) (N=22)
Constipation (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Tongue discomfort (Gastrointestinal disorders) | 0 | 1
Tongue erythema (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 1 | 1
Chest discomfort (General disorders) | 1 | 0
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Glucose urine present (Investigations) | 1 | 1
Glucose urine present (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Electrocardiogram ST segment elevation (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 0
Urine analysis abnormal (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 2
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT04511819/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT04511819/SAP_001.pdf